CLINICAL TRIAL: NCT02867852
Title: Phase II Trial of Abiraterone Acetate in Patients With Relapsed and/or Metastatic, Castration Resistant Salivary Gland Cancers
Brief Title: Abiraterone Acetate in Patients With Relapsed and/or Metastatic Salivary Gland Cancers
Acronym: SG-ABI14
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 71/14
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Salivary Glands Tumors
MeSH Terms: interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone acetate (Experimental): Abiraterone acetate 1 g/day must be taken as four 250-mg tablets daily on an empty stomach. No food should be consumed for at least 2 hours before the dose of abiraterone acetate is taken and for at least 1 hour after the dose of abiraterone acetate is taken. Prednisone (prednisolone when prednisone is not available) 5 mg will be given orally twice a day.
  Interventions: Drug: Abiraterone acetate

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone acetate is a prodrug of abiraterone, an irreversible inhibitor of 17α hydroxylase/C17, 20-lyase (cytochrome P450c17 [CYP17]), a key enzyme required for testosterone synthesis. This enzyme is found in the testes, adrenals, prostate tumors
  Other Names: Zytiga

SUMMARY:
Carcinomas of the salivary glands (SGCs) are rare tumors. Some selected salivary gland histotypes such as salivary duct carcinomas (SDC) and adenocarcinomas, NOS (not otherwise specified) distinguish themselves for the expression of androgen receptors (AR), which is reported in 21% to 43% of the cases. Thus, similarly to prostate cancer (Pca), androgen deprivation therapy (ADT) has been suggested to be beneficial in patients with recurrent or disseminated AR-expressing disease. No other therapy except palliative chemotherapy is available after progression on ADT, thus underling the necessity of alternative therapeutic approaches.

DETAILED DESCRIPTION:
Carcinomas of the salivary glands (SGC) are rare tumors. They comprise less than 1% of all cancers of the head and neck. The standard treatment is surgical excision, followed by radiotherapy in selected cases, such as high-grade tumors, and/or in the presence of perineural invasion, and/or in the presence of advanced disease. Some selected salivary gland histotypes such as salivary duct carcinomas (SDC) and adenocarcinomas, NOS (not otherwise specified) distinguish themselves for the expression of androgen receptors (AR), which is reported in 21% to 43% of the cases. Thus, similarly to prostate cancer (Pca), androgen deprivation therapy (ADT) has been suggested to be beneficial in patients with recurrent or disseminated AR-expressing disease.

The proven activity of ADT in AR expressing SGC as well as in Pca, suggests a common clinical behaviour by apparently sharing the same biological background. Once Pca becomes resistant to castration it still remains driven by ligand-dependent AR signaling and further hormonal manipulations are active and efficacious. Abiraterone acetate is currently approved by FDA for castration-resistant prostate cancer (CRPC). We treated with abiraterone two patients with AR-positive adenocarcinoma who had progressed on ADT, both patients showed a partial response suggesting the activity of a second line hormonal therapy in SGCs.

Based on the above biological and clinical evidences, the aim of the trial is to assess the activity of abiraterone in AR-expressing castration resistant SGCs.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥18 years
* Histologically or cytologically confirmed salivary glands cancer
* At least, one target lesion defined as RECIST 1.1 (clear progression of disease is required in the presence of one target lesion previously treated with radiotherapy
* Clinical and/or radiological progression of disease on ADT
* Ongoing androgen deprivation with a serum testosterone level of less than 50 ng per deciliter (1.7 nmol per liter)
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
* Adequate bone marrow function: Neutrophils > 1.5 x 109/L; Hemoglobin ≥ 9.0 g/dL independent of transfusion and platelet count ≥ 100,000/μL
* No limits are required for the number of previous chemotherapy lines
* Serum albumin ≥ 3.0 g/dL
* Serum creatinine <1.5 x upper limit of normal (ULN) or a calculated creatinine clearance ≥ 60 mL/min
* Serum potassium ≥3.5 mmol/L
* Able to swallow the study drug whole as a tablet
* Patients with treated brain metastases, stable within the last three months, are allowed
* Subjects who have partners of childbearing potential must use a method of birth control with adequate barrier protection as determined to be acceptable by the investigator and for 13 weeks after last study drug administration

Exclusion Criteria:

* Received abiraterone acetate within the last 5 years
* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Abnormal liver functions consisting of any of the following:
* Serum bilirubin ≥ 1.5 x ULN (except for subjects with documented Gilbert's disease, for whom the upper limit of serum bilirubin is 3 mg/dL)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2.5 x ULN
* Patients with ALT and/or AST not exceeding 5 x ULN due to liver mets can be enrolled
* Uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥95 mmHg); subjects with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive therapy
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease or left ventricular ejection fraction (LVEF) of <50% at baseline
* History of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study drug
* Any acute toxicities due to prior chemotherapy or radiotherapy that have not resolved to a NCI-CTCAE (Version 4.0) Grade of ≤1
* Participation in clinical trials with other experimental agents within 30 days of study entry or concomitant treatment with other experimental drug
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis and T1) or any cancer curatively treated > 3 years prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2019-11 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Response rate | 4 years
  The assessment of the activity considered as the response rate of abiraterone acetate in castration resistant salivary glands cancer

SECONDARY OUTCOMES:
Disease Control Rate | 4 years
  The assessment of disease control rate of abiraterone acetate in castration resistant salivary glands cancer
Adverse Events incidence | 4 years
  Incidence of adverse events, according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.0
Progression free survival | 4 years
  The assessment of progression free survival of patients suffering from castration resistant salivary glands cancer enrolled and treated wuth abiraterone acetate
Overall survival | 4 years
  The assessment of overall survival of patients suffering from castration resistant salivary glands cancer enrolled and treated wuth abiraterone acetate

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Licitra, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Abstract presentation to National and International congresses and final data publication on indexed papers

REFERENCES:
- [Derived] Locati LD, Cavalieri S, Bergamini C, Resteghini C, Colombo E, Calareso G, Mariani L, Quattrone P, Alfieri S, Bossi P, Platini F, Capone I, Licitra L. Abiraterone Acetate in Patients With Castration-Resistant, Androgen Receptor-Expressing Salivary Gland Cancer: A Phase II Trial. J Clin Oncol. 2021 Dec 20;39(36):4061-4068. doi: 10.1200/JCO.21.00468. Epub 2021 Oct 1. PMID 34597119